CLINICAL TRIAL: NCT01470586
Title: Surgical Resection Lowers Oxidative Stress Markers in Patients With Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. Hatzikosta General Hospital (Other)
Collaborators: University of Ioannina (Other)
Responsible Party: Principal Investigator, E.Tsimoyiannis, Head of Department of Surgery, G.Hatzikosta General Hospital, G. Hatzikosta General Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple
Other Study IDs: GH-1948-08
Record Dates: First submitted 2011-11-05; First posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Colorectal Cancer; Colon Rectal Resection; Oxidative Stress
Keywords: Colorectal cancer; Surgical resection; Oxidative Stress Markers; Controls
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgery for colorectal cancer (Other): Colorectal cancer patients
  Interventions: Procedure: Surgery for colorectal cancer
- Controls (No Intervention): Controls

INTERVENTIONS:
Procedure: Surgery for colorectal cancer — Surgical resection of colorectal cancer
  Other Names: Open or Laparoscopic resection for colorectal cancer; Low anterior resection; Sigmoidectomy; Left colectomy; Trasverse colectomy; Right colectomy
  Arms: Surgery for colorectal cancer

SUMMARY:
Study of Oxidative stress Markers (F2 Isoprostanes for lipid peroxidation, Carbonyl groups for protein peroxidation, 3 Nitrotyrosine for damage by nitrogens, and 8-Hydroxyguanosine for RNA peroxidation)in patients with colorectal cancer undergo surgical treatment (preoperatively during the intervention and postoperatively) and controls.

DETAILED DESCRIPTION:
Study of the impact of surgery on Lipid peroxidation, Protein peroxidation, damage by nitrogens, and RNA peroxidation, in patients undergo surgical resection for colorectal cancer and compared with controls, and validation of the responsiveness of oxidative stress markers on surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients with colorectal cancer
* Controls

Exclusion Criteria:

* ASA>3
* Metastatic Disease
* Acute bowel obstruction
* Acute bowel perforation
* BMI<30
* Chronic Systemic or Autoimmune Diseases
* Smokers
* Alcohol consumers

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Comparison of Oxidative stress markers in patients with colorectal cancer and controls | up to 2 years
  Oxidative stress markers variation (8-PGF2α, Protein Carboyls, 3-Nitrotyrosine, 8-OHG) during and after surgery for colorectal cancer, and compare with controls

SECONDARY OUTCOMES:
Validation of oxidative stress markers in patients with colorectal cancer undergo surgical resection | up to 2 years
  Validation of the responsiveness of markers of oxidative stress 8-PGF2α, Protein Carboyls, 3-Nitrotyrosine, 8-OHG)on surgery

CONTACTS AND LOCATIONS:
Overall Officials: George Pappas-Gogos, MD, Principal Investigator — G. Hatzikosta General Hospital
Locations (1):
- G. Hatzikosta General Hospital, Ioannina, Epirus, Greece